CLINICAL TRIAL: NCT05300620
Title: The Effect of Running Shoes With and Without Custom Foot Orthotics on Performance, Running Economy, Running Mechanics and Comfort
Brief Title: The Effect Custom Foot Orthotics on Comfort, Kinetics and Kinematics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspetar (Other)
Collaborators: Queen Margaret University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: F2017000201; REP0258 (Other: Queen Margaret Univeristy)
Record Dates: First submitted 2022-02-28; First posted 2022-03-29 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: Running economy; Orthotic Materials; Footwear comfort; Gait; Running

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Original Shoe Liner (Experimental): This condition will be administered by inserting the original liner in the shoe and have the participants run with this shoe condition.
  Interventions: Device: Original Liner
- Custom Foot Orthotic made out of Ethyl Vinyl Acetate material (Experimental): This condition will be administered by inserting a custom EVA orthotic in the shoe and have the participants run with this shoe condition.
  Interventions: Device: Custom Foot Orthotics EVA
- Custom Foot Orthotic made of thermoplastic poly-urethane material (Experimental): This condition will be administered by inserting a custom TPU orthotic in the shoe and have the participants run with this shoe condition.
  Interventions: Device: Custom Foot Orthotics PU
- Hybrid - Orthotic made of EVA and TPU material (Experimental): This condition will be administered by inserting a custom EVA/TPU orthotic in the shoe and have the participants run with this shoe condition.
  Interventions: Device: Custom Hybrid Foot Orthotics

INTERVENTIONS:
Device: Custom Foot Orthotics EVA — these are custom foot orthotics made out of Ethyl Vinyl Acetate material
  Arms: Custom Foot Orthotic made out of Ethyl Vinyl Acetate material
Device: Original Liner — these are original shoe liners
  Arms: Original Shoe Liner
Device: Custom Foot Orthotics PU — these are custom foot orthotics made out of Expanded Poly Urethane Material
  Arms: Custom Foot Orthotic made of thermoplastic poly-urethane material
Device: Custom Hybrid Foot Orthotics — these are custom foot orthotics made out of a combination of Ethyl Vinyl Acetate and Expanded Poly Urethane Material
  Arms: Hybrid - Orthotic made of EVA and TPU material

SUMMARY:
The overarching aim of this project is to investigate the role of custom foot orthotics in a 'return to performance' framework as the ultimate part of the 'return to sport continuum'.

The aim of this particular study is to investigate the effect of Custom Foot Orthotics (CFO) made from different materials on Running Economy (RE).

Well trained recreational athletes (volunteers) will present to a physiology lab for a familiarisation running session where standard measurements (e.g. height, weight, shoe size, training history, foot shape) will be recorded. During this initial visit, our volunteers will also perform an incremental running test to determine the individual ventilatory threshold (VT). This will allow the use of individual speeds of a relative equal intensity that which will be used during the experimental session. A full explanation of the experimental procedures will be given and trialed. This session will last about 1 hour.

For the experimental session (minimum of one week after the incremental test and receiving the custom-made orthotics), our volunteers will report to the same lab minimal 4 hours post prandial, having done no strenuous exercise for 12 hours before data collection. After a 10-minute warm up, Participants will run four 6-minute trials (four footwear conditions) with plenty of rest (5 minutes) between running trials to recover and answer short surveys on footwear comfort and readiness to start the next session.

Also actual sprint performance will be tested. After a 10-minute general and sprint specific warm up twelve 5-second all out sprints (3 sprints per condition) with 4 minutes recovery between each sprint will be performed.

This session will last about 2 and a half hours.

The volunteers will run in four different footwear conditions:

standardized running shoes + original liner of the sport shoe standardized running shoes + a custom-made orthotic from an EVA/TPU material standardized running shoes + a custom-made orthotic from an EVA material standardized running shoes + a custom-made orthotic from an TPU material

DETAILED DESCRIPTION:
Participants will attend the laboratory on two separate occasions. The first visit is to determine the individual ventilatory threshold (VT) and corresponding running speed that will be used for next intervention session by performing a VO2 max running test. The second visit will consist of running at submaximal speed in four different footwear conditions in randomized order, followed by three sprints in each different footwear condition in randomised order. Participants will run with standardized (i.e., only shoe liner inserted) footwear (Control), Standardised footwear with a Hybrid custom foot orthotic (Hybrid), Standardised footwear with an EVA custom foot orthotic (EVA) and Standardised footwear with a TPU custom foot orthotic (TPU) . Participants will be asked to avoid strenuous exercise in the 12 h, as well as refrain from food and caffeine for 4 h preceding their visits to the laboratory and are encouraged to replicate their diet and training pattern prior to all visits. Laboratory conditions will be monitored and kept similar throughout all running sessions. Furthermore, time of day will be standardized for each participant for both sessions. The participants and the researchers who will be directly involved in guiding the runners during the running protocol, and the statistical analysis are blinded from the exact footwear condition.

Running bouts

Visit 1 - Incremental test Each participant will complete a continuous, maximal incremental running test to determine their individual VT1 and according running speed. Briefly, participants start running at 9 km.h-1 for men and 7 km.h-1 for women with speed increases of 0.5 km.h-1 every 30 s. The test ends with voluntary exhaustion of the participants. Verbal encouragement will only be given by the researcher guiding the runners throughout the session.

Visit 2 - Sub-maximal runs and sprints After a ten-minute warm-up at a self-selected comfortable speed, followed by a 3-minute break used to put on the mask to collect expired gas, participants will run four, six-minute trials at a speed 10 % below VT speed, with five minutes recovery in between sessions.

During this time, each participant will

answer a survey regarding the comfort of their footwear. have their shoes removed and replaced by one of the researchers. answer a survey regarding their readiness to perform before starting the next 6-minute trial The order in which shoe conditions are applied will be randomized across participants and sessions (eg. steady state runs and sprint).

After the four submaximal runs participants will have a short break before starting the sprint sessions and warm up. After a 10-minute general and sprint specific warm up including a warmup run, stretching including hamstrings, 3 to 5 second accelerations with subjective increasing intensity of their perceived maximal effort, 3-second sprint at 80 and 90% of perceived maximal effort will be performed on the treadmill.

Twelve 5-second all-out sprints (3 sprints per footwear condition) will be performed. For the sprinting sessions, the participants will be attached with a rope around their waste that is tethered to an anker in the wall behind the treadmill. Participants will be required to lean forward in a typical and standardised crouched sprint-start position with their left foot forward (like in the picture above), which also will be explained, demonstrated, and tested during the first familiarisation session.

This starting position will be the same for all sprints. Participants will be guided with a 5-s countdown (eg. "5 s, 3-2-1-Go") given by both visual and audio instructions.

Between each 5 second sprint there will be 4 minutes recovery. During this recovery time, participants will

answer a survey regarding the comfort of their footwear. have their shoes removed and replaced by one of the researchers after each set of 3 sprints. (Participants will be able to lace their shoe to feel comfortable) answer a survey regarding their readiness to perform before starting the next sprint.

This session will last around approximately 2 and a half hours where you will be running and sprinting about 45 to 50 minutes. The rest of the time is used to prepare (eg. marker placement by researchers), recover and answer survey questions.

Footwear During all running the participants will use neutral like running shoes (Pearl Izumi N2v2, Colorado, US). With a minimum of seven days before the start of visit 2, each participant will receive three pairs of CFO based on an individual non-weight bearing 3D scan of the foot using an Elinvision iCube500 scanner (Elinvision, Karmėlava, Lithuania) that will be completed at the end of the first visit (incremental test). CFO will be designed by an experienced sports podiatrist with 20 years of experience, using FitFoot360 (Fit360 ltd, Worcestershire, UK). Briefly, scans will be imported into the software, markers placed over the heel, first- and fifth metatarsal and medial arch.

A base model surface shall be adjusted to match the contour of the foot using cross-sectional views from the heel to the forefoot. The thickness of the orthotic will be arbitrary set to 8 mm in an attempt to maximize the potential of the expanded thermoplastic polyrethane (TPU) beats inside the Infinergy® material (BASF, Ludwigshafen, Germany). All CFO are direct-milled out of a bespoke block of EVA on the rearfoot and TPU on the forefoot, a block of EVA and a block of TPU and manually finished to fit inside the shoes. The geometry of the supports will be exactly the same, only the material will be different.

On initial fitting and again before the start of the intervention session (second visit), participants will be asked if the CFO is comfortable and if any adjustments are necessary.

The weight of the four footwear conditions (shoe + liner or CFO) will also be recorded.

Data collection Instrumented treadmill An instrumented treadmill (ADAL3D-WR, Medical Developpement - HEF Techmachine, France) will be used for all running conditions (incremental test, steady-state running and sprint). Briefly, it is mounted on a highly rigid metal frame, set at 0˚ grade incline, fixed to the ground through four piezoelectric force transducers (KI 9077b; Kistler, Winterthur, Switzerland) and installed on a specially engineered concrete slab to ensure maximal rigidity of the supporting ground.

Metabolic card A Jeager™ Oxycon Mobile CPET unit (Carefusion, Hoechberg, Germany) will be to record breath-by-breath and cardio-respiratory data. Prior to each session, calibration of gas sensor is completed for ambient air and a known gas mixture (16 % O2, 5 % CO2). Turbine is calibrated using a 3-Liter (±0.4 %) syringe and automated High and Low flow ventilation. The metabolic cart is suspended from the ceiling next to participants, so Participants don't have to support the additional weight of the system when running.

Vicon Kinematic data will be collected using a modified Helen Hayes model utilizing 44 retroreflective markers fixed to the lower extremity skin. A static calibration trial to determine joint centers will be obtained utilizing medial anatomical markers. A three-dimensional motion capture system including thirteen cameras and Vicon Nexus Software (Vicon, Inc., Centennial, CO) will be used to capture at 200Hz, reduce, and analyse kinematic data. Using double-sided tape, the investigators will adhere small reflective markers bilaterally to the skin over: the ASIS and PSIS of the pelvis, the greater trochanter, the medial and lateral femoral condyles, and the medial and lateral malleoli. Markers are fixed to both shoes: one on the posterior of the heel, one below the medial and lateral malleolus, one each above the tips of the first and fourth toes, and one over the first and fifth metatarsal head. To track the movements of the thigh and shank segments which are assumed to be rigid bodies, plate marker sets consisting of a 4 marker cluster will be used. The plates will be attached to each thigh and calf segment using elastic bandage material.

ELIGIBILITY:
Inclusion Criteria:

* Well-trained (regularly running 35 km or more a week)

Exclusion Criteria:

* history of cardiovascular, neurological, or orthopaedic problems or musculoskeletal injury of the lower limb less than 3 months leading up to the data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in running economy | 16 times within the 2.5 hour session during the last 2 minutes of steady state running and sprint for each of the 4 footwear conditions
  VO2 per bodyweight over speed, expressed in milliliters of oxygen consumed per kilogram per kilometer using CPET.

SECONDARY OUTCOMES:
Change in Footwear Comfort | 16 times within the 2.5 hour session after each running bout
  (cushioning and control) and locations under the foot (heel, medial arch and forefoot) when compared to control (shoes only) using a standardised footwear comfort questionnaire ("the footwear comfort assessment tool" developed by Mundermann)
  Overall Comfort:
  What's the OVERALL impression of the insole COMFORT*
  Heel Cushioning:
  What's the impression of the softness/hardness of the HEEL REGION? *
  Forefoot Cushioning:
  What's the impression of the softness/hardness of the FOREFOOT REGION? *
  Overall Control:
  What's the OVERALL impression of the orthotic in CONTROLLING THE POSITION of your foot? *
  Medial Arch Height What's the impression of the push you feel in the ARCH on the inside of your feet? *
  Heel Cup Fit What's the impression on the FIT of the insole ie. whether the insole is loose or tight? *
  *For each section a score can be given between 0 = Not comfortable at all 150 = most comfortable condition imaginable Higher scores means better outcome
Change in running kinetics | 16 times within the 2.5 hour session during the last 2 minutes of steady state running and sprint for each of the 4 footwear conditions
  Three-dimensional Force related measure using ADAL instrumented treadmill, measured in Newtons.
change in running kinematics | 16 times within the 2.5 hour session during the last 2 minutes of steady state running and sprint for each of the 4 footwear conditions
  Three-dimensional Movement related measure, using VICON motion capture measured in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Marco Cardinale, Prof, Study Director — Aspetar Orthopeadic and Sports Medicine Hospital
Locations (1):
- Aspetar, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Alsenoy K, Ryu JH, Girard O. The Effect of EVA and TPU Custom Foot Orthoses on Running Economy, Running Mechanics, and Comfort. Front Sports Act Living. 2019 Sep 19;1:34. doi: 10.3389/fspor.2019.00034. eCollection 2019. PMID 33344957
- [Background] Girard O, Morin JB, Ryu JH, Van Alsenoy K. Custom foot orthoses improve performance, but do not modify the biomechanical manifestation of fatigue, during repeated treadmill sprints. Eur J Appl Physiol. 2020 Sep;120(9):2037-2045. doi: 10.1007/s00421-020-04427-0. Epub 2020 Jun 30. PMID 32607818